CLINICAL TRIAL: NCT01512771
Title: The Effect of Nasal Continuous Positive Airway Pressure (Nasal CPAP) Treatment on Post Traumatic Stress Disorder (PTSD) Symptoms.
Brief Title: The Effect of Nasal Continuous Positive Airway Pressure Treatment on PTSD Symptoms.
Acronym: PTSD
Status: Completed | Type: Observational
Sponsor: Northport Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mohammad M Amin, Staff Physician, Northport Veterans Affairs Medical Center
Other Study IDs: 00383
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Post Traumatic Stress Disorder; Anxiety; Nightmares; Unrefreshed Sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: CPAP — 6 weeks of CPAP

SUMMARY:
We hypothesize that prevention of Sleep Disordered Breathing among PTSD patients with nasal CPAP will result improve their anxiety, insomnia and alcohol craving (among those who use alcohol to control their symptoms).

DETAILED DESCRIPTION:
Design: This is a pilot study to study the effect of nasal CPAP on the symptoms of PTSD in veterans.

Recruitment Methods:

Veterans with PTSD will be recruited from the Northport VAMC PTSD unit. The ACOS/Mental Health will refer patients that meet inclusion criteria and do not have an impaired decision making capacity. Subjects will be screened for decision-making capacity by their treating psychiatrist as part of their clinical assessment upon admission to the PTSD unit.

Study Methods

This will be a prospective, randomized, controlled interventional trial:

1. Participants will undergo a routine clinical sleep study at the PTSD unit (using a portable polysomnographic recording unit). or undergo a routine clinical polysomnography to diagnose sleep disordered breathing
2. Participants who demonstrate SDB will be randomized into two groups based upon their body mass index

   1. Group A: BMI < 30 kg/m2
   2. Group B: BMI > 30 kg/m2 The reason for these two arms is to study the effect of nasal CPAP upon PTSD symptoms in veterans with a high prevalence of sleep apnea ( BMI above 30 kg/m2) and in veterans with predominantly snoring (BMI below 30 kg/m2).

   Each group will then be randomized into two sub-groups regarding treatment.
   1. Treatment group receives an automated CPAP unit to use during sleep for 6 weeks in conjunction with their usual care in the PTSD unit (psychotherapy).
   2. Control group receives the usual care that is provided in the PTSD unit for 6 weeks (change in medications will exclude the subject from the study), if any participant in the control group would like to try nasal CPAP, then he will be crossed over to use an automated CPAP unit during sleep for his second 6 weeks in the PTSD unit together with usual care.
3. All participants will fill out the following questionnaires at baseline and after 6 weeks. (Those in the control group who have been crossed-over to nasal CPAP will also fill out a set of questionnaire at 12 weeks).

   1. PTSD checklist-military version (anxiety)
   2. MASQ anxious arousal subscale (anxiety)
   3. Insomnia Severity Index (insomnia)
   4. The alcohol craving questionnaire (with an alcohol history during the intake) The changes in patient's reported outcomes will be compared before and after CPAP treatment and psychotherapy alone

ELIGIBILITY:
Inclusion Criteria:

A. Admitted to PTSD unit at NVAMC and will remain in the unit for at least 12 weeks after initiation of study participation.

B. Found to have SDB by polysomnography

Exclusion Criteria:

1. Impaired Decision-Making Capacity, as determined by treating psychiatrist.
2. No sleep disordered breathing found by polysomnography
3. Unable/unwilling to use the nasal CPAP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: veterans admitted to PTSD unit at Northport VAMC
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The Effect of nasal Continuous Positive Airway Pressure (nasal CPAP) Treatment on Post Traumatic Stress Disorder (PTSD) Symptoms. | six weeks of nasal CPAP
  A comparison of the effectiveness of six weeks of nasal CPAP plus usual care to usual care alone at decreasing the symptoms of PTSD (anxiety, insomnia and alcohol craving) among veterans with PTSD and SDB

SECONDARY OUTCOMES:
The Effect of nasal Continuous Positive Airway Pressure (nasal CPAP) Treatment on Post Traumatic Stress Disorder (PTSD) Symptoms. | 6 weeks of nasal CPAP
  A comparison of the change in symptoms to the change in the total of sleep stage shifts during sleep for all patients with PTSD and SDB participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Amin, MD, Principal Investigator — Northport VAMC
Locations (1):
- PTSD unit at Northport VAMC, Northport, New York, United States